CLINICAL TRIAL: NCT01648270
Title: Influence of Cyclosporine on Buprenorphine Disposition
Brief Title: Buprenorphine Disposition and Cyclosporine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201202087
Record Dates: First submitted 2012-04-10; First posted 2012-07-24 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: buprenorphine; CYP3A
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Subjects will be studied on four occasions. Sessions and drugs are:
  1. Intravenous buprenorphine
  2. Sublingual buprenorphine
  3. Cyclosporine plus intravenous buprenorphine
  4. Cyclosporine plus sublingual buprenorphine
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — Session 1 Intravenous buprenorphine: 0.2 mg over 1 hr Session 2 Sublingual buprenorphine: 2 mg Session 3 Intravenous buprenorphine 0.2 mg over 1 hr beginning 1 hr after starting cyclosporine Session 4 Sublingual buprenorphine: 2 mg after cyclosporine.

SUMMARY:
The determine the effect of cyclosporine on buprenorphine disposition

DETAILED DESCRIPTION:
Subjects studied on four occasions:

1. Intravenous buprenorphine
2. Sublingual buprenorphine
3. Cyclosporine, then intravenous buprenorphine. Subjects then take oral cyclosporine twice daily, until
4. Sublingual buprenorphine; continue oral cyclosporine twice daily for 5 days

ELIGIBILITY:
Inclusion Criteria:

* 18-50 yr old
* Good general health with no remarkable medical conditions
* BMI < 33
* Provide informed consent

Exclusion Criteria:

* Known history of liver or kidney disease
* Use of prescription or non prescription medications, herbals or foods known to be metabolized by or affecting CYP3A
* Females who are pregnant or nursing
* Known history of drug or alcohol addiction (prior or present addiction or treatment for addiction)
* Direct physical access to and routine handling of addicting drugs in the regular course of duty (a routine exclusion from studies of drugs with addiction potential)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine: Subjects will be studied on four occasions. Sessions and drugs are:
  1. Intravenous buprenorphine
  2. Sublingual buprenorphine
  3. Cyclosporine plus intravenous buprenorphine
  4. Cyclosporine plus sublingual buprenorphine
Period: Intravenous Buprenorphine
Arm/Group | Buprenorphine
Started | 25
Completed | 13
Not Completed | 12
Not completed — Withdrawal by Subject | 12
Period: Sublingual Buprenorphine
Arm/Group | Buprenorphine
Started | 13
Completed | 13
Not Completed | 0
Period: Cyclosporine Plus IV Buprenorphine
Arm/Group | Buprenorphine
Started | 13
Completed | 13
Not Completed | 0
Period: Cyclosporine + Sublingual Buprenorphine
Arm/Group | Buprenorphine
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Plasma Cmax
Time Frame: 96 hours
Population: 0 Participants Analyzed. The PI has left the institution. Sincere efforts were made to contact the PI but were unsuccessful. No study data are available.
Groups:
- Intravenous Buprenorphine: Intravenous buprenorphine: 0.2 mg infused over 1 hr
- Sublingual Buprenorphine: Sublingual buprenorphine: 2 mg
- Cyclosporine + IV Buprenorphine: Cyclosporine (2.5mg/kg/hr infused over 2 hr), then intravenous buprenor-phine 0.2 mg infused over 1 hr beginning 1 hr after starting cyclosporine. Subjects then take oral cyclosporine 4.5 mg/kg twice daily
- Cyclosporine + Sublingual Buprenorphine: Sublingual buprenorphine: 2 mg; continue oral cyclosporine 4.5 mg/kg twice daily for 5 days
Arm/Group | Intravenous Buprenorphine | Sublingual Buprenorphine | Cyclosporine + IV Buprenorphine | Cyclosporine + Sublingual Buprenorphine
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Groups:
- Cyclosporine Plus Intravenous Buprenorphine: Cyclosporine (2.5mg/kg/hr infused over 2 hr), then intravenous buprenor-phine 0.2 mg infused over 1 hr beginning 1 hr after starting cyclosporine. Subjects then take oral cyclosporine 4.5 mg/kg twice daily
- Cyclosporine Plus Sublingual Buprenorphine: Sublingual buprenorphine: 2 mg; continue oral cyclosporine 4.5 mg/kg twice daily for 5 days
Arm/Group | Intravenous Buprenorphine | Sublingual Buprenorphine | Cyclosporine Plus Intravenous Buprenorphine | Cyclosporine Plus Sublingual Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 16/18 | 17/18 | 17/18 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Buprenorphine (N=18) | Sublingual Buprenorphine (N=18) | Cyclosporine Plus Intravenous Buprenorphine (N=18) | Cyclosporine Plus Sublingual Buprenorphine (N=18)
nausea (Gastrointestinal disorders) | 10 (10) | 13 (13) | 10 (10) | 9 (9)
itch (General disorders) | 12 (12) | 14 (14) | 8 (8) | 11 (11)
Headache (Nervous system disorders) | 6 (6) | 3 (3) | 2 (2) | 4 (4)
Dizzyness (Nervous system disorders) | 4 (4) | 5 (5) | 3 (3) | 1 (1)
Other (Product Issues) | 2 (2) | 1 (1) | 10 (10) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes